CLINICAL TRIAL: NCT05427942
Title: YUflyma® (Adalimumab), Patient Experience After Switching to adaliMumab biosimilAr High concenTration, Low Volume (40mg/0.4mL) (Yuflyma®) by Taking Patient pERception of Treatment Into Account: The YU-MATTER Study
Brief Title: Yuflyma® (Adalimumab), Patient Experience After Switching
Acronym: YU-MATTER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Celltrion HealthCare France (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022-A00448-35
Record Dates: First submitted 2022-06-17; First posted 2022-06-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Rheumatoid Arthritis; Ankylosing Spondylarthritis; Axial Spondyloarthritis Without Radiographic Evidence of Ankylosing Spondylitis; Psoriatic Arthritis; Crohn Disease; Ulcerative Colitis
Keywords: CT-P17; Patient experience; Satisfaction; Biosimilar
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylitis, Ankylosing; Non-Radiographic Axial Spondyloarthritis; Arthritis, Psoriatic; Crohn Disease; Colitis, Ulcerative; Personal Satisfaction | interventions — Adalimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Switch from adalimumab originator
  Interventions: Drug: Adalimumab
- Switch from adalimumab biosimilar 40 mg/0,8 mL
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Adalimumab — Stable and treated for at least 3 months prior to inclusion either with an adalimumab biosimilar or originator adalimumab (40 mg dose injections only) and for whom the treating physician has decided to switch to Yuflyma® (40 mg / 0.4 mL) on the day of their inclusion (decision independent from the study)

SUMMARY:
Patient preference and experience can impact patients' adherence and persistence regarding a treatment, especially when switching. A number of factors contribute to this, including their beliefs, fears, expectations, and overall knowledge. This is compounded by the fact that many switched patients are not trained on how to use the new injection device.

Specifically, some patients report a degraded experience with current adalimumab biosimilars (40mg/0.8mL) as compared to the originator: injections appear more painful and seem to cause more bruising. Indeed, treatment-related factors such as treatment volume or the presence of citrate have the potential to negatively impact patient experience and contribute to local reactions at or around the injection site, such as pain and swelling.

Yuflyma® (CT-P17 adalimumab), developed by Celltrion Inc., is a biosimilar of the anti-TNF treatment adalimumab, having obtained a marketing authorisation from the European Commission on 11th February 2021 (addressed to Celltrion Healthcare).

Yuflyma® is the first high-concentration adalimumab biosimilar (40mg/0.4mL) available in France, which makes the product similar to the currently available adalimumab originator formula in terms of drug concentration.

Studying patient experience over the course of a switch involves querying patients at the time of prescription, while they are still under the previous treatment, and for the following 3 months, during which they have been able to pick up their prescribed medication from a pharmacy and have started using the new treatment. Describing patient experience over the course of a switch from another adalimumab (originator or biosimilar) to Yuflyma® would contribute to identifying significant factors which contribute to patient experience and satisfaction.

Our primary objective is to assess patients' overall satisfaction with the injection after the switch to the high-concentration adalimumab biosimilar Yuflyma®, at 3 months following the initiation, compared to their experience with the previous adalimumab.

* Overall satisfaction with the injection (7-level likert) before initiation
* Overall satisfaction with the injection (7-level likert) 3 months after initiation

ELIGIBILITY:
Inclusion Criteria:

* Adult (aged 18 or older at the time of inclusion) rheumatology or gastroenterology patients presenting a diagnosis for any of the following pathologies : Rheumatoid Arthritis (RA) Ankylosing Spondylarthritis (AS) Axial Spondyloarthritis with no signs of AS (AxSpa) Psoriatic Arthritis (PsA) Crohn's Disease (CD) Ulcerative Colitis (UC)
* Stable and treated for at least 3 months prior to inclusion either with an adalimumab (ADA) biosimilar or originator adalimumab (40 mg dose injections only)
* For whom the treating physician has decided to switch to Yuflyma® (40 mg / 0.4 mL) on the day of their inclusion (decision independent from the study)
* Able to initiate treatment within 4 weeks of inclusion
* Have an email account
* Have a mobile phone number
* Able to understand and complete French-language questionnaires
* Are not opposed to participating in the study.
* Are covered by French National Health Insurance.

Non inclusion Criteria:

Patients meeting any of the following exclusion criteria will not be included in the study:

* Patients younger than 18 years old at the date of inclusion
* Patients treated with adalimumab for any other pathology than those specified in the inclusion criteria.
* Patients treated with adalimumab originator 80 mg.
* Patients under curatorship or guardianship or otherwise deprived of liberty
* Patients unable to understand and complete French-language questionnaires
* Pregnant women or women of childbearing potential with a desire of becoming pregnant concomitant to treatment with Yuflyma®.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult rheumatology or gastroenterology patients presenting a diagnosis for any of the following pathologies:
  * Rheumatoid Arthritis (RA)
  * Ankylosing Spondylarthritis (AS)
  * Axial Spondyloarthritis with no signs of AS (AxSpa)
  * Psoriatic Arthritis (PsA)
  * Crohn's Disease (CD)
  * Ulcerative Colitis (UC) Participants are included by practising physicians.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-06-03 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Overall satisfaction | March 2023
  Assess patients' overall satisfaction with the injection after the switch to the high-concentration adalimumab biosimilar Yuflyma®, at 3 months following the initiation, compared to their experience with the previous adalimumab.
  * Overall satisfaction with the injection (7-level likert) before initiation
  * Overall satisfaction with the injection (7-level likert) 3 months after initiation

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Private Practice - ES, Marseille
  - Private practice GB, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bouguen G, Gossec L, Abitbol V, Senbel E, Bonnaud G, Roblin X, Bouhnik Y, Nancey S, Mathieu N, Filippi J, Vuitton L, Nahon S, Dellal A, Denis A, Foulley L, Habauzit C, Benkhalifa S, Marotte H. Patient Satisfaction and Experience with CT-P17 Following Transition from Reference Adalimumab or Another Adalimumab Biosimilar: Results from the Real-World YU-MATTER Study. BioDrugs. 2024 Nov;38(6):867-878. doi: 10.1007/s40259-024-00681-2. Epub 2024 Sep 25. PMID 39322802
- See also: eCRF platform — https://yu-matter.sanoia.com